CLINICAL TRIAL: NCT00140634
Title: Cartilage Repair Registry
Brief Title: The Objectives of the Cartilage Repair Registry is to Report Long Term Efficacy and Safety of Cartilage Repair Procedures in Registry Patients
Status: Completed | Type: Observational
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Cartilage Repair Registry
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Articular Cartilage; Cartilage Diseases
MeSH Terms: conditions — Cartilage Diseases | interventions — Drug Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Carticel (autologous cultured chondrocyte) implantation — Each Carticel vial of autologous cultured chondrocytes contains approximately 12 million cells implanted into the defect and secured with a periosteal flap.

SUMMARY:
The objectives of the Cartilage Repair Registry is to report the long term efficacy and safety of cartilage repair procedures in Registry patients.

ELIGIBILITY:
Inclusion Criteria:

* All registry patients meeting the cohort definition at the pre-operative visit will be included on the overall summary tables for the patient cohort

Exclusion Criteria:

* All registry patients meeting the cohort definition at the pre-operative visit will be included on the overall summary tables for the patient cohort

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Registry of patients with diagnosis of chondral injury.
Sampling Method: Non-Probability Sample
Enrollment: 2233 (Actual)
Dates: Start 1995-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Physician assessment of effectiveness of autologous chondrocyte implantation | 6 month post implantation
  Overall assessment of the patient by the physician based on knee examination and progress of rehabilitation
Physician assessment of effectiveness of autologous chondrocyte implantation | 12 month post implantation
  Overall assessment of the patient by the physician based on knee examination and progress of rehabilitation
Physician assessment of effectiveness of autologous chondrocyte implantation | 24 month post implantation
  Overall assessment of the patient by the physician based on knee examination and progress of rehabilitation

SECONDARY OUTCOMES:
Patient assessment of effectiveness of autologous chondrocyte implantation | 6 month post implantation
  Overall assessment of the patient by the patient based on pain, swelling, giving-way, grinding, stiffness, catching and locking and quantity of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Registry contains data from patients whom were implanted by 1123 surgeons in the U.S. and also data captured on patients treated by 154 surgeons in 15 other countries., Cambridge, Massachusetts, United States